CLINICAL TRIAL: NCT02689635
Title: The Salt Trial: Low Sodium vs. Regular Diet in Patients Admitted for Heart Failure
Brief Title: Low Sodium vs. Regular Diet in Patients Admitted for Heart Failure
Acronym: SALT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI transferred to a new institution
Sponsor: Maya Guglin (Other)
Responsible Party: Sponsor-Investigator, Maya Guglin, Professor, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-0387-F3R
Record Dates: First submitted 2016-02-05; First posted 2016-02-24 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Diet, Sodium-Restricted; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Restricted Diet (Active Comparator): Low Salt (cardiac) diet
  Interventions: Other: Sodium Restricted Diet
- Regular Diet (Active Comparator): Non-Cardiac diet
  Interventions: Other: Regular Diet

INTERVENTIONS:
Other: Sodium Restricted Diet — Cardiac Diet, as defined by our Hospital Nutritional Services (containing less than 2000 mg sodium per day)
  Arms: Sodium Restricted Diet
Other: Regular Diet — Non-Cardiac Diet, as defined by our Hospital Nutritional Services
  Arms: Regular Diet

SUMMARY:
Patients over 18 years of age, admitted to the hospital with HF exacerbation, will be eligible for randomization to low salt or regular diet. Laboratory tests are routinely obtained on admission and on the day (or the day before) of discharge (comprehensive metabolic panel and NT-proBNP) and will be recorded for the study. Daily weights are routinely recorded, and intake/output will be monitored. At discharge, a Diet Acceptability Questionnaire will be performed.

After the discharge, participants will return for follow-up visits as needed for clinical indications. Our study coordinator will document changes of symptoms, changes in therapies, and capture clinical events like unscheduled hospital visits or visits to the Emergency Room. Once during the study patients will be asked about their specific food consumption on a prior day, and the Sodium content will be estimated. The final visit will occur in a year (approximately 11-13 months after enrollment). Weight, other vital signs, CMP, BNP, and Diet Acceptability Questionnaire quality of life questionnaire will be collected at this point, if clinically indicated.

The majority of study information will be collected from routine care for standard clinical indications. The only components added for study purpose are Diet Acceptability Questionnaire and collection of the information on consumed foods.

DETAILED DESCRIPTION:
This study will include patients over 18 years of age, admitted to the hospital with HF exacerbation, will be eligible for randomization to low salt or regular diet. Laboratory tests are routinely obtained on admission and on the day (or the day before) of discharge (comprehensive metabolic panel and NT-proBNP) and will be recorded for the study. Daily weights are routinely recorded, and intake/output will be monitored. At discharge, a Diet Acceptability Questionnaire will be performed.

After the discharge, participants will return for follow-up visits as needed for clinical indications. Our study coordinator will document changes of symptoms, changes in therapies, and capture clinical events like unscheduled hospital visits or visits to the Emergency Room. Once during the study patients will be asked about their specific food consumption on a prior day, and the Sodium content will be estimated. The final visit will occur in a year (approximately 11-13 months after enrollment). Weight, other vital signs, CMP, BNP, and Diet Acceptability Questionnaire quality of life questionnaire will be collected at this point, if clinically indicated.

The majority of study information will be collected from routine care for standard clinical indications. The only components added for study purpose are Diet Acceptability Questionnaire and collection of the information on consumed foods.The number of total days in the hospital for heart failure throughout the year will be compared between the arms.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Hospital admission for principal diagnosis of heart failure
* Left ventricular ejection fraction </=40%

Exclusion Criteria:

* Concomitant hypertension (blood pressure >150/90 mmHg on admission and at least twice more during the index stay)
* Planned LVAD or Heart Transplant in next 3 months
* Patient on current or planned renal dialysis
* Inability to give the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Readmission Rate | 12 months
  Number of hospital and ER admissions during the 1 year follow up period

SECONDARY OUTCOMES:
Length of stay | from time of hospital admission to hospital discharge, up to one year
  number of days hospitalized
Total length of stay | 1 year follow up period
  total days admitted to hospital during follow up period
Weight | measured daily during hospital admission period, up to one year
NT-pro BNP, pg/mL | at the time of hospital admission and time of hospital discharge, up to one year
Diet Satisfaction as assessed by the Diet Acceptability Questionnaire | at the time of hospital discharge (final hospitalization day, up to one year) and one year

CONTACTS AND LOCATIONS:
Overall Officials: Maya Guglin, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No